CLINICAL TRIAL: NCT04133194
Title: Adherence of a 1.600 mg Single Tablet 5-ASA Treatment of Ulcerative Colitis (EASI-trial)
Brief Title: Adherence of a 1.600 mg Single Tablet 5-ASA Treatment of Ulcerative Colitis
Acronym: EASI
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Flemming Bendtsen (Other)
Responsible Party: Sponsor-Investigator, Flemming Bendtsen, Professor, Senior doctor, MDSci, Copenhagen University Hospital, Hvidovre
Organization: Copenhagen University Hospital, Hvidovre (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1337-EASI-trial
Record Dates: First submitted 2019-10-10; First posted 2019-10-21 (Actual); Last update posted 2023-09-26 (Actual); Status verified 2023-09

CONDITIONS: Ulcerative Colitis
MeSH Terms: conditions — Colitis, Ulcerative | interventions — Mesalamine

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- 1600 mg Asacol (mesalazine) (Experimental): 1600 mg mesalazine (Asacol) treatment regimen (1 tablet per day) for a year
  Interventions: Drug: Mesalazine
- 800 mg Asacol (mesalazine) (Active Comparator): 800 mg mesalazine (Asacol) treatment regimen (3 tablets per day) for a year
  Interventions: Drug: Mesalazine

INTERVENTIONS:
Drug: Mesalazine — 1600 mg Asacol [mesalazine]
  Arms: 1600 mg Asacol (mesalazine)
Drug: Mesalazine — 800 mg Asacol [mesalazine]
  Arms: 800 mg Asacol (mesalazine)

SUMMARY:
Several oral mesalazine (5-ASA) formulations exist, but the regimes require several tablets per day. Such regimens are not ideal and can interfere with normal daily activities of patients. Non-adherence has been associated with an increase in the risk of relapse and worse disease course; leading to a decrease in quality of life, an increase in societal and personal costs, and worst case increases the risk of colorectal cancer. Recently, a new formula for 5-ASA has been approved by the Danish Medicine Agency, with a single tablet regime per day.

Primary purpose:

• To investigate whether a simplified treatment regimen for 5- ASA (1600 mg as one tablet per day [intervention]) improves adherence with preserved remission rates compared to conventional therapy.

Secondary purposes:

* Compare levels of endoscopic, mucosal and histological inflammation in predicting risk of relapse between the intervention group and the conventional therapy group.
* Investigate whether a simplified treatment regimen improves the disease course compared to the conventional therapy.
* To assess the correlation between different endpoints and the disease courses, with the use of clinical, endoscopic, histological, self-reported and biochemical markers.
* Improve, correlate and assess patient-reported outcomes in a prospective manner.
* To establish a biobank of cases with quiescent/mild ulcerative colitis (UC) for identification of future biomarkers.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent
* Age between and including 18 and 60
* Diagnosed with UC according to the Copenhagen Diagnostic Criteria
* Length of disease of max. 10 years
* Stable remission on 5-ASA (defined as partial Mayo score ≤1) for at least 2 months without need for oral corticosteroids before inclusion.
* Endoscopic remission defined as Mayo Clinic Endoscopic Score < 2
* Have had a relapse within the last 2 years

  * Defined as the need of escalation of treatment or change medical treatment.

Exclusion Criteria:

* Evidence of infectious diarrhoea (i.e. pathogenic viruses, bacteria or Clostridium difficile toxin in stool culture) within the last month
* On immunomodulators, including methotrexate
* On any biological therapy
* Any previous abdominal surgery related to UC
* Any chronic infections (e.g. HBV, HCV, HIV)
* Any severe concomitant cardiovascular, autoimmune, hematologic, hepatic, renal, endocrine, oncologic or psychiatric disorder, which in the opinion of the investigator might have an influence on the patient's compliance or the interpretation of the results
* Well-founded doubt about the patient's cooperation, e.g., because of addiction to alcohol or drugs in the opinion of the investigators.
* Participation in another clinical trial within the last 30 days, or simultaneous participation in another clinical trial.
* Any previous documented allergic reaction to tested the medical drugs

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 200 (Estimated)
Dates: Start 2019-11-28 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-03-01 (Estimated)

PRIMARY OUTCOMES:
Medical Adherence | through study completion, an average of 2 year
  Measured by drug accountability log
  Patients having taken ≥80 % are categorised as adherent
Medical Adherence | through study completion, an average of 2 year
  Measured by "Medical adherence rating scale" (MARS)
  Medical adherence rating scale is a self-reported medical adherence tool consisting of 5 items scored on a 5 point Likert scale (ranging from 5-25). The scale has been used in several IBD studies and a global score > 20 indicates a good adherence.
Medical Adherence | through study completion, an average of 2 year
  Measured byf drug accountability log (outcome 1) and "Medical adherence rating scale" (MARS, outcome 2) separately, excl. pregnant and breastfeeding women.
  Further detail see outcome 1 and 2

SECONDARY OUTCOMES:
Assessment of disease activity by Mayo Score | through study completion, an average of 2 year
  The Mayo Score is composed of 4 items. A score from 0-2 is categorised as remission and 11-12 as severe.
Assessment of disease activity by the Simple clinical colitis activity index (SCCAI) | through study completion, an average of 2 year
  The SCCAI rely solely on clinical assessments. Clinical remission are defined as SCCAI < 1 and clinical response as a change of at least 1 point.
Assessment of endoscopic severity by the Ulcerative Colitis Endoscopic Index of Severity (UCEIS) | through study completion, an average of 2 year
  The UCEIS endoscopic severity on a scale of 1-4. Higher score mean worse disease severity.
Assessment of endoscopic severity by the Mayo endoscopic score | through study completion, an average of 2 year
  The Mayo endoscopic score is scored on a scale of 0-3. Higher score mean worse disease severity.
Assessment of histological severity by the Geboes score | through study completion, an average of 2 year
  The Geboes score is interpreted as such: a higher score means higher disease activity.
Assessment of histological severity by the Nancy Index | through study completion, an average of 2 year
  The Nancy Index are interpreted as such: The grade 4 correspond to severe disease, grade 0 as " absence of significant histological disease".
Assessment of histological severity by the Robarts Histopathology Index (RHI) | through study completion, an average of 2 year
  The RHI are interpreted as such: The score are ranging between 0 (no disease activity) to 33 (severe disease activity).
Correlation between the different clinical scores | through study completion, an average of 2 year
  Comparison, correlation and association between the different endoscopic, histological and disease activity indices.
  Included will be:
  Mayo score, Simple clinical colitis activity index (SCCAI), Ulcerative Colitis Endoscopic Index of Severity (UCEIS), Nancy Index, Robarts Histopathology Index (RHI) and the Geboes score (see outcome 4-10).
Remission - days | through study completion, an average of 2 year
  Differences in number of days in remission during the trial
Relapse - days | through study completion, an average of 2 year
  Differences in number of days in relapse during the trial
Remission and relapse - episodes | through study completion, an average of 2 year
  Differences episodes of relapses during the trial
Changes in quality of life | through study completion, an average of 2 year
  Prospective analyses of quality of life using 12-Item Short Form Survey (SF12).
  The SF12 is measured on a global score from 12-56. Beside a global score, a mental and physical dimension will also be calculated.
Changes in disease specific quality of life | through study completion, an average of 2 year
  Prospective analyses quality of life using the Short inflammatory bowel disease questionnaire (SIBDQ)
  The SIBDQ is a quality of life (QOL) questionnaire ranging from 10-70. Higher score means better QOL.
Changes in disability among ulcerative colitis patients | through study completion, an average of 2 year
  Prospective analyses of disability using the Inflammatory bowel disease disability index (IBD-DI)
  The IBD-DI measures the disability among patients with inflammatory bowel disease. Higher scores means worse disability.
Changes in sleep quality | through study completion, an average of 2 year
  Prospective analyses of sleep using the Pittsburgh Sleep Quality Index (PSQI),
  The PSQI was designed to measure sleep quality and disturbance. A global score > 5 is considered poor sleep quality.
Changes in resilience | through study completion, an average of 2 year
  Prospective analyses of resilience using the Brief Resilience Scale (BRS)
  The BRS is designed to measure the ability to bounce back or recover from stressful events. Higher scores means higher resilience.

CONTACTS AND LOCATIONS:
Overall Officials: Flemming Bendtsen, MDSci, Principal Investigator — Copenhagen University Hospital, Hvidovre
Locations (1):
- Copenhagen University Hospital Hvidovre, Hvidovre, Denmark

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR

REFERENCES:
- [Derived] Nordestgaard RLM, Lo B, Bergstrom R, Adzioski I, Skotte H, Hawwa IM, Holme SK, Tiftikci B, Majchrzak K, Vind I, Bendtsen F, Burisch J. Clinical Trial: Evaluating a Single 1600 mg Tablet Regimen of 5-Aminosalicylate for Ulcerative Colitis-The EASI Trial. Aliment Pharmacol Ther. 2025 Nov;62(9):877-886. doi: 10.1111/apt.70375. Epub 2025 Sep 16. PMID 40955556